CLINICAL TRIAL: NCT06287190
Title: Assessment of Self-Confidence of Dental Interns Regarding Provision of Different Pediatric Dentistry Procedures: A Before and After Study
Brief Title: Assessment of Self-Confidence of Dental Interns Regarding Provision of Different Pediatric Dentistry Procedures
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Laila Khalid H. Halawani, Principal Investigator, Doctor Laila Halawani, Cairo University
Other Study IDs: Self-confidence assessment
Record Dates: First submitted 2024-02-12; First posted 2024-03-01 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Self Confidence
Keywords: dental interns; pediatric dentistry; assessment; treatment

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dental interns: Assessing dental intern confidence before and after finishing their rotation at the pediatric department
  Interventions: Other: Dental interns

INTERVENTIONS:
Other: Dental interns — Assessing self-assessment

SUMMARY:
This study mainly about dental interns testing their knowledge before and after entering the pediatric rotation

DETAILED DESCRIPTION:
A convenient sample will be selected from the dental interns attending the Pediatric Dentistry Department, Cairo University training period. The study will include all the dental interns submitted for training over 12 successive months.

ELIGIBILITY:
Inclusion Criteria:

* Dental interns who got their bachelor's degree from Egyptian governmental and private universities.
* Dental interns who passed the internship period in the pediatric dentistry department.

Exclusion Criteria:

* Dental interns who got their bachelor's degrees from abroad universities.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Dental interns who are taking their internship at the Cairo university
Sampling Method: Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Self-confidence regarding treatment | during first month
  Questionnaire regarding self confidence

SECONDARY OUTCOMES:
difficulties in dental practice through this period | up to 12 months
  Questionnaire about the difficulties

CONTACTS AND LOCATIONS:
Overall Officials: Sherine E Eldin, Prof, Study Chair — Professor in Pediatric Dentistry and Public Health Department Faculty of Dentistry, Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yiu CK, McGrath C, Bridges S, Corbet EF, Botelho MG, Dyson JE, Chan LK. Self-perceived preparedness for dental practice amongst graduates of The University of Hong Kong's integrated PBL dental curriculum. Eur J Dent Educ. 2012 Feb;16(1):e96-e105. doi: 10.1111/j.1600-0579.2011.00681.x. Epub 2011 Feb 17. PMID 22251360
- [Result] Togoo R, Nasim V, Zakirulla M, Yaseen S. Knowledge and Practice of Pulp Therapy in Deciduous Teeth among General Dental Practitioners in Saudi Arabia. Ann Med Health Sci Res. 2012 Jul;2(2):119-23. doi: 10.4103/2141-9248.105657. PMID 23440030
- [Result] Shelton A, Yepes JF, Vinson LA, Jones JE, Tang Q, Eckert GJ, Downey T, Maupome G. Utilization of Stainless Steel Crowns by Pediatric and General Dentists. Pediatr Dent. 2019 Mar 15;41(2):127-131. PMID 30992110
- [Result] Rodd HD, Farman M, Albadri S, Mackie IC. Undergraduate experience and self-assessed confidence in paediatric dentistry: comparison of three UK dental schools. Br Dent J. 2010 Mar 13;208(5):221-5. doi: 10.1038/sj.bdj.2010.207. PMID 20228757
- [Result] SWY, Wong & XQ, Wong & Vaithilingam, Rathna & Rajan, Sadna. (2015). Dental Undergraduates' Self-Assessed Confidence in Paediatric Dentistry. Annals of Dentistry. 22. 9. 10.22452/adum.vol22no2.4
- See also: elf-assessed Confidence of Dentists in Pediatric Dentistry: A cross-sectional study — http://pjmhsonline.com/index.php/pjmhs/article/view/19